CLINICAL TRIAL: NCT02627365
Title: Motivation Matters! Randomized Clinical Trial of Theory Based SMS to Support Treatment as Prevention in High-Risk Women
Brief Title: Motivation Matters Study
Acronym: MM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Nairobi (Other); Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Scott McClelland, Professor, Medicine, Epidemiology, and Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00000394
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: HIV/AIDS
Keywords: ART; mobile messaging; behaviour; motivation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individualized, interactive SMS (Experimental): Individualized, interactive SMS intervention plus Standard care. Messages sent automatically using the Text-IT system.
  Interventions: Behavioral: Individualized, interactive short messaging intervention
- Standard care (No Intervention): Standard care according to Kenyan guidelines, including clinic-based adherence education and counseling.

INTERVENTIONS:
Behavioral: Individualized, interactive short messaging intervention — An Individualized, interactive short messaging intervention reminding study participants to take antiretroviral medication and report any problems.
  Arms: Individualized, interactive SMS

SUMMARY:
The study aims to develop and evaluate the efficacy and causal mechanisms of an interactive SMS intervention to optimize individual health and secondary HIV prevention benefits of ART in HIV-positive FSWs.

DETAILED DESCRIPTION:
Antiretroviral therapy (ART) is highly effective at reducing the infectiousness of HIV-positive people, and is considered the cornerstone of all new HIV prevention approaches. A critical question is how to harness the potency of ART to reduce transmission from female sex workers (FSWs), a key population that has been central to HIV transmission in Africa for more than 25 years. In high prevalence countries like Kenya, FSWs represent about 1% of the population, yet contribute to one in seven (14%) new HIV infections. Targeting treatment as prevention (TasP) to FSWs could efficiently reduce HIV transmission on a population level. Effective TasP will require higher levels of ART adherence than those achieved in typical treatment programs. The rapid spread of mobile technology in Africa provides unique opportunities for mobile health (mHealth) interventions, which have been shown to be acceptable to providers and patients, and can improve ART adherence and suppression of plasma HIV viral load.

The ability of mobile (SMS) interventions to support ART adherence in key populations like FSWs and unique clinical scenarios such as TasP has yet to be evaluated. The investigators will answer these fundamental questions by addressing the following aims: 1) To use a qualitative rapid assessment and development approach to craft a theory-based, individualized, interactive SMS intervention, grounded in the Theory of Information, Motivation, and Behavior (IMB), to support ART adherence in HIV-positive FSWs, 2) To compare individualized, interactive SMS to standard care in achieving undetectable HIV VL 6 months post ART initiation in a randomized controlled trial (RCT) with 210 FSWs and 3) To administer an adaptation of the LifeWindows Information - Motivation - Behavioral Skills ART Adherence Questionnaire (LW-IMB-AAQ) to understand the mechanism of our SMS intervention's effect by comparing perceptions of support and motivation to adhere to ART in FSWs who received the intervention versus standard care.

Our overarching goal is to develop and evaluate the efficacy and causal mechanisms of an interactive SMS intervention to optimize individual health and secondary HIV prevention benefits of ART in HIV-positive FSWs. The aims of this project proceed sequentially from developmental (Aim 1) through implementation of the intervention (Aim 2) to evaluation of the fit with the behavioral model (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years or emancipated minor
* Has access to mobile phone
* Self-identifying female sex worker
* Willing to receive study SMS messages
* HIV-positive (any WHO stage or CD4)
* Able to read or have someone else read
* ART naïve
* Informed consent obtained and signed.

Exclusion Criteria:

* Plans to move away in next 6 months
* Contraindication to ART

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2016-01; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Plasma HIV-1 viral load | six months
  The plasma HIV-1 viral load will be compared between participants in the intervention and in the non-intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: R. Scott McClelland, M.D, MPH, Principal Investigator — University of Washington
Locations (1):
- Women's Health Project, Mombasa, Mombasa, Kenya

REFERENCES:
- [Derived] Aunon FM, Wanje G, Richardson BA, Masese L, Odeny TA, Kinuthia J, Mandaliya K, Jaoko W, Simoni JM, McClelland RS. Randomized controlled trial of a theory-informed mHealth intervention to support ART adherence and viral suppression among women with HIV in Mombasa, Kenya: preliminary efficacy and participant-level feasibility and acceptability. BMC Public Health. 2023 May 8;23(1):837. doi: 10.1186/s12889-023-15638-3. PMID 37158872
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730